CLINICAL TRIAL: NCT04298385
Title: A Non-Invasive and Low-Profile Dynamic Traction Orthosis for Oblique Proximal Phalangeal Fractures: A Case Series
Brief Title: Traction Orthosis for Oblique Proximal Phalangeal Fractures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southern Health and Social Care Trust (Other Government)
Responsible Party: Principal Investigator, Daniel Harte, Advanced Occupational Therapist, Southern Health and Social Care Trust
Other Study IDs: V4 20012020
Record Dates: First submitted 2020-01-30; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Trauma; Fractures, Bone; Finger Fracture
MeSH Terms: conditions — Wounds and Injuries; Fractures, Bone | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with oblique proximal phalanx fractures of finger: Traction orthosis and exercise
  Interventions: Other: Traction orthosis

INTERVENTIONS:
Other: Traction orthosis — Traction applied to a finger using elastic thread and sports tape and attached to an orthosis
  Other Names: exercise

SUMMARY:
The term Ligamentotaxis is used to define the method of distal traction to realign joint surfaces and reduce articular fragments after complex fractures.

Traction and mobilization can be combined to help deliver the best outcome.

This study will present a dynamic traction orthosis design with the aim that it is easy-to-make, non-invasive, low-profile and allow for ease in performing active and passive exercises. The clinical effectiveness of this method will be examined by analyzing treatment outcomes in a case series cohort.

DETAILED DESCRIPTION:
The term Ligamentotaxis is used to define the method of distal traction to realign joint surfaces and reduce articular fragments after complex fractures. In the management of complex finger fractures, ligamentotaxis has been used to favourably help fracture alignment and reduction, range of movement (ROM), pain, grip and function. Traction has been applied via nail anchors skin traction and Kirschner wires.

Phalangeal fractures are at risk of chronic stiffness when immobilised. Early mobilization seeks to achieve the best outcome for the patient as it will aid healing, promote cartilage regeneration, help prevent adhesions and optimize range of movement. Mobilisation of phalangeal fractures as soon as possible after open reduction internal fixation has shown to produce greater total range of movement at six weeks post-operatively. Traction and mobilization can be combined to help deliver the best outcome however dynamic traction orthoses tend to be "high-profile". This can cause difficulties in activities of daily living and can be perceived negatively by users. Most dynamic traction orthoses use Kirschner wires which have the potential complication of loosening and pin site infection.

Two methods report good outcomes using the less invasive and less expensive means of tape and nail traction respectively. The Early Active Vector Adjustable Skin Traction (EAVAST) orthosis has no reported issues using adhesive tape though the patient is required to remove the orthosis to perform exercises. This removes any stability offered by the orthosis during the early phases of healing. The Poole traction orthosis is well-established in some centres with reported good outcomes however nail traction has the potential complication of nail bed haematoma or nail avulsion.

A recent orthosis design by the Chief Investigator aspired to be non-invasive, low-profile and allow for ease when performing exercises. However, this design may be deemed too time consuming to make, particularly for the inexperienced therapist in a busy clinic. This study will present a further iteration of the dynamic traction orthosis with the aim that it is easy-to-make, non-invasive, low-profile and allow for ease in performing active and passive exercises. The clinical effectiveness of this method will be examined by analyzing treatment outcomes in a case series cohort.

The new orthosis design will be easy to fabricate and can be produced with common materials and tools in a hand therapy clinic. It offers a non-invasive approach to dynamic traction and simultaneously is easy to perform a variety of tendon glides and active and passive exercises. It also reduces the risk associated with nail traction and pinning. It is low-profile ensuring range of motion is maintained in non-affected joints and helps participation in activities of daily living. The proposed case series will illustrate this method and explore its clinical application by presenting outcomes.

Though a recent scoping review reports that research addressing traction orthoses and constructs consists of primarily low-quality studies and no consensus on the their effect on different fracture classifications, this small study will act as a feasibility study to assess the orthosis design with a focus on displaced oblique proximal phalangeal fractures or potentially unstable oblique proximally phalangeal fractures

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years and over who are able to provide informed consent and independently comply with the orthosis and exercise regime
* A recent oblique proximal phalangeal fracture that is displaced or has the potential to become unstable. The decision for trial of a dynamic traction orthosis must be made by the orthopaedic surgeon
* No history of trauma or disease to the affected hand

Exclusion Criteria:

* A fracture which is more than 10 days from injury

  * An open wound around the affected digit
  * A history of allergic reactions to plasters
  * Eczema or dermatitis to the affected hand
  * The presence of sensory loss to the affected digit
  * Ligament or tendon injury that will contra-indicate early mobilisation
  * Transverse proximal phalanx fractures
  * A tattoo to the affected hand that may prevent anonymity when producing photographs

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People who have sustained a recent oblique proximal phalanx fractures that is displaced or potentially unstable
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Range of motion | up to three months post intervention
  Goniometer: Measures in degrees range of movement of a joint
Pain and function | up to three months post intervention
  Patient Related Wrist Hand Evaluation: a Likert scale that measure pain and function on a total score of 0-100
Grip | up to three months post intervention
  Dynamometer: measure hand grip in Ibs and can be compared to normative data

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schenck RR. Dynamic traction and early passive movement for fractures of the proximal interphalangeal joint. J Hand Surg Am. 1986 Nov;11(6):850-8. doi: 10.1016/s0363-5023(86)80236-2. PMID 3794242
- [Result] Collins AL, Timlin M, Thornes B, O'Sullivan T. Old principles revisited--traction splinting for closed proximal phalangeal fractures. Injury. 2002 Apr;33(3):235-7. doi: 10.1016/s0020-1383(01)00138-3. PMID 12084639
- [Result] Fitzgerald JA, Khan MA. The conservative management of fractures of the shafts of the phalanges of the fingers by combined traction-splintage. J Hand Surg Br. 1984 Oct;9(3):303-6. doi: 10.1016/0266-7681(84)90048-2. PMID 6512368
- [Result] Goldman SB, Amaker RJ, Espinosa RA. James traction splinting for PIP fractures. J Hand Ther. 2008 Apr-Jun;21(2):209-15. doi: 10.1197/j.jht.2007.08.019. PMID 18436143
- [Result] Jehan S, Chandraprakasam T, Thambiraj S. Management of proximal phalangeal fractures of the hand using finger nail traction and a digital splint: a prospective study of 43 cases. Clin Orthop Surg. 2012 Jun;4(2):156-62. doi: 10.4055/cios.2012.4.2.156. Epub 2012 May 17. PMID 22662302
- [Result] Baier S, Szekeres M. The hand arc--a hand-based splint design for intraarticular fractures. J Hand Ther. 2010 Jan-Mar;23(1):73-76. doi: 10.1016/j.jht.2009.07.006. Epub 2009 Nov 1. PMID 19883994
- [Result] Byrne A, Yau T. A modified dynamic traction splint for unstable intra-articular fractures of the proximal interphalangeal joint. J Hand Ther. 1995 Jul-Sep;8(3):216-8. doi: 10.1016/s0894-1130(12)80022-6. No abstract available. PMID 8535487
- [Result] Kadelbach D. Swing design dynamic traction splinting for the treatment of intra-articular fractures of the digits. J Hand Ther. 2006 Jan-Mar;19(1):39-42. doi: 10.1197/j.jht.2005.11.001. PMID 16473733
- [Result] Murray KA, McIntyre FH. Active traction splinting for proximal interphalangeal joint injuries. Ann Plast Surg. 1995 Jul;35(1):15-8. doi: 10.1097/00000637-199507000-00003. PMID 7574279
- [Result] Hardy MA. Principles of metacarpal and phalangeal fracture management: a review of rehabilitation concepts. J Orthop Sports Phys Ther. 2004 Dec;34(12):781-99. doi: 10.2519/jospt.2004.34.12.781. PMID 15643733
- [Result] Feehan LM, Bassett K. Is there evidence for early mobilization following an extraarticular hand fracture? J Hand Ther. 2004 Apr-Jun;17(2):300-8. doi: 10.1197/j.jht.2004.02.014. PMID 15162112
- [Result] Chinchalkar SJ, Gan BS. Management of proximal interphalangeal joint fractures and dislocations. J Hand Ther. 2003 Apr-Jun;16(2):117-28. doi: 10.1016/s0894-1130(03)80007-8. PMID 12755163
- [Result] Miller L, Ada L, Crosbie J, Wajon A. Pattern of recovery after open reduction and internal fixation of proximal phalangeal fractures in the finger: a prospective longitudinal study. J Hand Surg Eur Vol. 2017 Feb;42(2):137-143. doi: 10.1177/1753193416670591. Epub 2016 Oct 4. PMID 27702779
- [Result] O'Brien L, Presnell S. Patient experience of distraction splinting for complex finger fracture dislocations. J Hand Ther. 2010 Jul-Sep;23(3):249-9; quiz 260. doi: 10.1016/j.jht.2010.01.002. PMID 20399606
- [Result] Packham TL, Ball PD, MacDermid JC, Bain JR, DalCin A. A scoping review of applications and outcomes of traction orthoses and constructs for the management of intra-articular fractures and fracture dislocations in the hand. J Hand Ther. 2016 Jul-Sep;29(3):246-68. doi: 10.1016/j.jht.2016.04.001. PMID 27496982
- [Result] Spurrier E, Pathak G, Khanna A. Pressure exerted by finger traps. J Perioper Pract. 2011 Apr;21(4):140-1. doi: 10.1177/175045891102100405. PMID 21560555
- [Result] Mathiowetz V, Kashman N, Volland G, Weber K, Dowe M, Rogers S. Grip and pinch strength: normative data for adults. Arch Phys Med Rehabil. 1985 Feb;66(2):69-74. PMID 3970660